CLINICAL TRIAL: NCT04515095
Title: A Safety and Feasibility Study of Water-only Fasting and Refeeding for Treatment of Stage 1 and 2 Hypertensive Patients
Brief Title: Water-only Fasting in the Treatment of Hypertension Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TrueNorth Health Foundation (Other)
Responsible Party: Principal Investigator, Toshia Myers, Director, TrueNorth Health Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNHF2020-1HTN
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hypertension
Keywords: fasting; water-only fasting; whole-plant-food diet
MeSH Terms: conditions — Hypertension; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Water-only Fasting Group (Experimental): Participants who voluntarily elect and are approved to water-only fast.
  Interventions: Other: Water-only Fasting

INTERVENTIONS:
Other: Water-only Fasting — Participants consume only water for at least 7 days in an in-patient, residential setting with 24 hour medical supervision.

SUMMARY:
This purpose of this study is to examine the safety and feasibility of water-only fasting to treat hypertensive patients.

DETAILED DESCRIPTION:
This is a prospective, open label, single arm, intervention study to examine the safety and feasibility of water-only fasting to treat hypertensive patients. Additional aims include describing mean changes in resting blood pressure as well as markers of cardiovascular health and inflammation between baseline and end of fast, end of refeed, 6-weeks post departure, and 12-months after 6-weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender
2. 30-75 years old
3. Diagnosis of Stage 1 or 2 hypertension
4. Fasting plasma glucose <126mg/dL and/or hemoglobin A1c <7 percent
5. Elect and qualify for a water-only fast of at least 7 consecutive days
6. Provide informed consent
7. Internet and computer access
8. Able to go to LabCorp for 6-week follow-up visit
9. Willing/able to collect 24-hour urine sample prior to water-only fasting

Exclusion Criteria:

1. Systolic Blood Pressure/Diastolic Blood Pressure >180/120 mmHg
2. Active malignancy
3. Active kidney disease (creatinine over 2.0)
4. Active inflammatory disorder including classic autoimmune connective tissue (Lupus, Sjogrens, ANCA), multiple sclerosis, and inflammatory bowel disorders (Ulcerative colitis, Crohn's)
5. Stroke, heart attack, deep vein thrombosis, atrial fibrillation, anticoagulant therapy, or pulmonary embolism within the last 12 months
6. Inability to discontinue medications or supplements
7. Abdominal metal implants
8. Inability to consume only plant food for at least 48 hours before fast begins.
9. Unable to lay still on the back for at least 10 min.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-16 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Determine number of treatment-associated of grade 1-4 adverse events as assessed by CTCAE v5.0 | up to 10-60 days after baseline
  Adverse events will be identified through participant interviews and medical record review

SECONDARY OUTCOMES:
Examine the feasibility of using fasting and refeeding in the treatment of stage 1 and 2 hypertension based on change in systolic blood pressure (SBP) | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast, 6-weeks after departure, 12-months after 6-weeks follow-up
  SBP will be measured using digital blood pressure device and reported in mmHg
Examine the feasibility of using fasting and refeeding in the treatment of stage 1 and 2 hypertension based on treatment acceptability | Up to 7-40 days after baseline and 6-weeks after end of refeed
  Treatment acceptability will be assessed using the validated Treatment Adherence/Acceptability Questionnaire
Examine the feasibility of using fasting and refeeding in the treatment of stage 1 and 2 hypertension based on food acceptability | 6-weeks after end of refeed
  Food acceptability will be assed using the validated Food Acceptability Questionnaire
Examine the feasibility of using fasting and refeeding in the treatment of stage 1 and 2 hypertension based on dietary adhernece | 6-weeks after end of refeed
  Dietary adherence rates will be assessed using the SOS-free Dietary Screener

OTHER OUTCOMES:
Describe mean changes in resting blood pressure from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in SBP and diastolic blood pressure will be measured using a digital blood pressure device and reported as mmHg
Describe mean changes in lipid profile from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in lipid profile will be assessed using serum to measure cholesterol, triglycerides, high-density lipoprotein (HDL), and low-density lipoprotein (LDL) and reported in mg/dL
Describe mean changes in fasting glucose and apolipoprotein B from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in fasting glucose and apolipoprotein B will be assessed using serum and reported as mg/dL
Describe mean changes in body mass index (BMI) from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in BMI will be assessed by measuring weight in kilograms (kg) and height in meters (m) and reported as kg/m2
Describe mean changes in insulin from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in insulin will be assessed by using serum and reported as uIU/ml
Describe mean changes in visceral adipose tissue from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed
  Changes in visceral adipose tissue will be assessed using dual-energy X-ray absorptiometry and presented as grams
Describe mean changes in high sensitivity C-reactive protein (hsCRP) from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in hsCRP will be assessed using serum and reported as mg/L
Describe mean changes in gamma-glutamyl-transferase (GGT) from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in GGT will be assessed using serum and reported as U/L
Describe mean changes in lipoprotein associated phospholipase A2 from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in lipoprotein associated phospholipase A2 will be assessed using serum and reported as nmol/min/mL
Describe mean changes in homocysteine from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in homocysteine will be assessed using serum and reported as umol/L
Describe mean changes in aldosterone from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in aldosterone will be assessed using serum and 24 hour urine and reported as ng/dL
Describe mean changes in abdominal circumference from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Abdominal circumference will be measured at minimal waist and reported in centimeters
Describe changes in renin activity from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in renin activity will be assessed using serum and reported as ng/mL/hr
Describe changes in sodium from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in sodium will be assessed using 24 hour urine and reported as mmol/24 hr
Describe changes in creatinine and total protein from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in sodium will be assessed using 24 hour urine and reported as mg/dL
Describe changes in potassium from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in potassium will be assessed using 24 hour urine and reported as mmol/L
Describe changes in albumin from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed, 12-months after 6-weeks follow-up
  Changes in albumin will be assessed using 24 hour urine and reported as ug/mL
Describe changes in 3-methyl-histidine from baseline | Baseline, up to 7-40 days after baseline, up to 3 to 20 days after end-of-fast, 6-weeks after end of refeed
  Changes in 3-methyl-histidine will be assessed using 24 hour urine and reported as umol/day

CONTACTS AND LOCATIONS:
Overall Officials: Toshia R Myers, PhD, Principal Investigator — Director
Locations (1):
- TrueNorth Health Center, Santa Rosa, California, United States

IPD SHARING:
Plan to Share IPD: Yes
After publication, the IPD will be available by contacting the corresponding author.

REFERENCES:
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Rapsomaniki E, Timmis A, George J, Pujades-Rodriguez M, Shah AD, Denaxas S, White IR, Caulfield MJ, Deanfield JE, Smeeth L, Williams B, Hingorani A, Hemingway H. Blood pressure and incidence of twelve cardiovascular diseases: lifetime risks, healthy life-years lost, and age-specific associations in 1.25 million people. Lancet. 2014 May 31;383(9932):1899-911. doi: 10.1016/S0140-6736(14)60685-1. PMID 24881994
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2018 May 15;71(19):e127-e248. doi: 10.1016/j.jacc.2017.11.006. Epub 2017 Nov 13. No abstract available. PMID 29146535
- [Background] Chockalingam A, Campbell NR, Fodor JG. Worldwide epidemic of hypertension. Can J Cardiol. 2006 May 15;22(7):553-5. doi: 10.1016/s0828-282x(06)70275-6. PMID 16755308
- [Background] Franklin SS. Ageing and hypertension: the assessment of blood pressure indices in predicting coronary heart disease. J Hypertens Suppl. 1999 Dec;17(5):S29-36. PMID 10706323
- [Background] Wall HK, Hannan JA, Wright JS. Patients with undiagnosed hypertension: hiding in plain sight. JAMA. 2014 Nov 19;312(19):1973-4. doi: 10.1001/jama.2014.15388. No abstract available. PMID 25399269
- [Background] Lawes CM, Bennett DA, Feigin VL, Rodgers A. Blood pressure and stroke: an overview of published reviews. Stroke. 2004 Apr;35(4):1024. PMID 15053002
- [Background] Forouzanfar MH, Liu P, Roth GA, Ng M, Biryukov S, Marczak L, Alexander L, Estep K, Hassen Abate K, Akinyemiju TF, Ali R, Alvis-Guzman N, Azzopardi P, Banerjee A, Barnighausen T, Basu A, Bekele T, Bennett DA, Biadgilign S, Catala-Lopez F, Feigin VL, Fernandes JC, Fischer F, Gebru AA, Gona P, Gupta R, Hankey GJ, Jonas JB, Judd SE, Khang YH, Khosravi A, Kim YJ, Kimokoti RW, Kokubo Y, Kolte D, Lopez A, Lotufo PA, Malekzadeh R, Melaku YA, Mensah GA, Misganaw A, Mokdad AH, Moran AE, Nawaz H, Neal B, Ngalesoni FN, Ohkubo T, Pourmalek F, Rafay A, Rai RK, Rojas-Rueda D, Sampson UK, Santos IS, Sawhney M, Schutte AE, Sepanlou SG, Shifa GT, Shiue I, Tedla BA, Thrift AG, Tonelli M, Truelsen T, Tsilimparis N, Ukwaja KN, Uthman OA, Vasankari T, Venketasubramanian N, Vlassov VV, Vos T, Westerman R, Yan LL, Yano Y, Yonemoto N, Zaki ME, Murray CJ. Global Burden of Hypertension and Systolic Blood Pressure of at Least 110 to 115 mm Hg, 1990-2015. JAMA. 2017 Jan 10;317(2):165-182. doi: 10.1001/jama.2016.19043. PMID 28097354
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] Kirkland EB, Heincelman M, Bishu KG, Schumann SO, Schreiner A, Axon RN, Mauldin PD, Moran WP. Trends in Healthcare Expenditures Among US Adults With Hypertension: National Estimates, 2003-2014. J Am Heart Assoc. 2018 May 30;7(11):e008731. doi: 10.1161/JAHA.118.008731. PMID 29848493
- [Background] Heidenreich PA, Trogdon JG, Khavjou OA, Butler J, Dracup K, Ezekowitz MD, Finkelstein EA, Hong Y, Johnston SC, Khera A, Lloyd-Jones DM, Nelson SA, Nichol G, Orenstein D, Wilson PW, Woo YJ; American Heart Association Advocacy Coordinating Committee; Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Arteriosclerosis; Thrombosis and Vascular Biology; Council on Cardiopulmonary; Critical Care; Perioperative and Resuscitation; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease; Council on Cardiovascular Surgery and Anesthesia, and Interdisciplinary Council on Quality of Care and Outcomes Research. Forecasting the future of cardiovascular disease in the United States: a policy statement from the American Heart Association. Circulation. 2011 Mar 1;123(8):933-44. doi: 10.1161/CIR.0b013e31820a55f5. Epub 2011 Jan 24. PMID 21262990
- [Background] Ames MK, Atkins CE, Pitt B. The renin-angiotensin-aldosterone system and its suppression. J Vet Intern Med. 2019 Mar;33(2):363-382. doi: 10.1111/jvim.15454. Epub 2019 Feb 26. PMID 30806496
- [Background] Buglioni A, Cannone V, Sangaralingham SJ, Heublein DM, Scott CG, Bailey KR, Rodeheffer RJ, Sarzani R, Burnett JC. Aldosterone Predicts Cardiovascular, Renal, and Metabolic Disease in the General Community: A 4-Year Follow-Up. J Am Heart Assoc. 2015 Dec 23;4(12):e002505. doi: 10.1161/JAHA.115.002505. PMID 26702078
- [Background] Cannone V, Buglioni A, Sangaralingham SJ, Scott C, Bailey KR, Rodeheffer R, Redfield MM, Sarzani R, Burnett JC Jr. Aldosterone, Hypertension, and Antihypertensive Therapy: Insights From a General Population. Mayo Clin Proc. 2018 Aug;93(8):980-990. doi: 10.1016/j.mayocp.2018.05.027. PMID 30077215
- [Background] Dudenbostel T, Calhoun DA. Use of Aldosterone Antagonists for Treatment of Uncontrolled Resistant Hypertension. Am J Hypertens. 2017 Feb;30(2):103-109. doi: 10.1093/ajh/hpw105. Epub 2016 Sep 8. PMID 27609503
- [Background] Bronsert MR, Henderson WG, Valuck R, Hosokawa P, Hammermeister K. Comparative effectiveness of antihypertensive therapeutic classes and treatment strategies in the initiation of therapy in primary care patients: a Distributed Ambulatory Research in Therapeutics Network (DARTNet) study. J Am Board Fam Med. 2013 Sep-Oct;26(5):529-38. doi: 10.3122/jabfm.2013.05.130048. PMID 24004705
- [Background] Wright JM, Musini VM, Gill R. First-line drugs for hypertension. Cochrane Database Syst Rev. 2018 Apr 18;4(4):CD001841. doi: 10.1002/14651858.CD001841.pub3. PMID 29667175
- [Background] Gebreyohannes EA, Bhagavathula AS, Abebe TB, Tefera YG, Abegaz TM. Adverse effects and non-adherence to antihypertensive medications in University of Gondar Comprehensive Specialized Hospital. Clin Hypertens. 2019 Jan 15;25:1. doi: 10.1186/s40885-018-0104-6. eCollection 2019. PMID 30675379
- [Background] Gupta R, Guptha S. Strategies for initial management of hypertension. Indian J Med Res. 2010 Nov;132(5):531-42. PMID 21150005
- [Background] Siervo M, Lara J, Chowdhury S, Ashor A, Oggioni C, Mathers JC. Effects of the Dietary Approach to Stop Hypertension (DASH) diet on cardiovascular risk factors: a systematic review and meta-analysis. Br J Nutr. 2015 Jan 14;113(1):1-15. doi: 10.1017/S0007114514003341. Epub 2014 Nov 28. PMID 25430608
- [Background] Chiavaroli L, Viguiliouk E, Nishi SK, Blanco Mejia S, Rahelic D, Kahleova H, Salas-Salvado J, Kendall CW, Sievenpiper JL. DASH Dietary Pattern and Cardiometabolic Outcomes: An Umbrella Review of Systematic Reviews and Meta-Analyses. Nutrients. 2019 Feb 5;11(2):338. doi: 10.3390/nu11020338. PMID 30764511
- [Background] Grillo A, Salvi L, Coruzzi P, Salvi P, Parati G. Sodium Intake and Hypertension. Nutrients. 2019 Aug 21;11(9):1970. doi: 10.3390/nu11091970. PMID 31438636
- [Background] McDougall J, Thomas LE, McDougall C, Moloney G, Saul B, Finnell JS, Richardson K, Petersen KM. Effects of 7 days on an ad libitum low-fat vegan diet: the McDougall Program cohort. Nutr J. 2014 Oct 14;13:99. doi: 10.1186/1475-2891-13-99. PMID 25311617
- [Background] McDougall J, Thomas LE, McDougall C, Moloney G, Saul B, Finnell JS, Richardson K, Petersen KM. Erratum to: Effects of 7 days on an ad libitum low-fat vegan diet: the McDougall Program cohort. Nutr J. 2017 Feb 10;16(1):12. doi: 10.1186/s12937-017-0234-9. No abstract available. PMID 28187767
- [Background] Huang L, Trieu K, Yoshimura S, Neal B, Woodward M, Campbell NRC, Li Q, Lackland DT, Leung AA, Anderson CAM, MacGregor GA, He FJ. Effect of dose and duration of reduction in dietary sodium on blood pressure levels: systematic review and meta-analysis of randomised trials. BMJ. 2020 Feb 24;368:m315. doi: 10.1136/bmj.m315. PMID 32094151
- [Background] Beauchesne AB, Goldhamer AC, Myers TR. Exclusively plant, whole-food diet for polypharmacy due to persistent atrial fibrillation, ischaemic cardiomyopathy, hyperlipidaemia and hypertension in an octogenarian. BMJ Case Rep. 2018 Dec 17;11(1):e227059. doi: 10.1136/bcr-2018-227059. PMID 30567282
- [Background] Tuso PJ, Ismail MH, Ha BP, Bartolotto C. Nutritional update for physicians: plant-based diets. Perm J. 2013 Spring;17(2):61-6. doi: 10.7812/TPP/12-085. PMID 23704846
- [Background] Esselstyn CB. A plant-based diet and coronary artery disease: a mandate for effective therapy. J Geriatr Cardiol. 2017 May;14(5):317-320. doi: 10.11909/j.issn.1671-5411.2017.05.004. No abstract available. PMID 28630609
- [Background] Goldhamer A, Lisle D, Parpia B, Anderson SV, Campbell TC. Medically supervised water-only fasting in the treatment of hypertension. J Manipulative Physiol Ther. 2001 Jun;24(5):335-9. doi: 10.1067/mmt.2001.115263. PMID 11416824
- [Background] Finnell JS, Saul BC, Goldhamer AC, Myers TR. Is fasting safe? A chart review of adverse events during medically supervised, water-only fasting. BMC Complement Altern Med. 2018 Feb 20;18(1):67. doi: 10.1186/s12906-018-2136-6. PMID 29458369
- [Background] Tchkonia T, Thomou T, Zhu Y, Karagiannides I, Pothoulakis C, Jensen MD, Kirkland JL. Mechanisms and metabolic implications of regional differences among fat depots. Cell Metab. 2013 May 7;17(5):644-656. doi: 10.1016/j.cmet.2013.03.008. Epub 2013 Apr 11. PMID 23583168
- [Background] Pepys MB, Hirschfield GM. C-reactive protein: a critical update. J Clin Invest. 2003 Jun;111(12):1805-12. doi: 10.1172/JCI18921. No abstract available. PMID 12813013
- [Background] Ganguly P, Alam SF. Role of homocysteine in the development of cardiovascular disease. Nutr J. 2015 Jan 10;14:6. doi: 10.1186/1475-2891-14-6. PMID 25577237
- [Background] Kumar A, Palfrey HA, Pathak R, Kadowitz PJ, Gettys TW, Murthy SN. The metabolism and significance of homocysteine in nutrition and health. Nutr Metab (Lond). 2017 Dec 22;14:78. doi: 10.1186/s12986-017-0233-z. eCollection 2017. PMID 29299040
- [Background] Mann NJ, Li D, Sinclair AJ, Dudman NP, Guo XW, Elsworth GR, Wilson AK, Kelly FD. The effect of diet on plasma homocysteine concentrations in healthy male subjects. Eur J Clin Nutr. 1999 Nov;53(11):895-9. doi: 10.1038/sj.ejcn.1600874. PMID 10557004
- [Background] Gilstrap LG, Wang TJ. Biomarkers and cardiovascular risk assessment for primary prevention: an update. Clin Chem. 2012 Jan;58(1):72-82. doi: 10.1373/clinchem.2011.165712. Epub 2011 Nov 28. PMID 22125305
- [Background] Tiu SC, Choi CH, Shek CC, Ng YW, Chan FK, Ng CM, Kong AP. The use of aldosterone-renin ratio as a diagnostic test for primary hyperaldosteronism and its test characteristics under different conditions of blood sampling. J Clin Endocrinol Metab. 2005 Jan;90(1):72-8. doi: 10.1210/jc.2004-1149. Epub 2004 Oct 13. PMID 15483077
- [Background] Stock J. Triglycerides and cardiovascular risk: Apolipoprotein B holds the key. Atherosclerosis. 2019 May;284:221-222. doi: 10.1016/j.atherosclerosis.2019.03.004. Epub 2019 Mar 21. No abstract available. PMID 30914143
- [Background] Ference BA, Kastelein JJP, Catapano AL. Lipids and Lipoproteins in 2020. JAMA. 2020 Aug 11;324(6):595-596. doi: 10.1001/jama.2020.5685. No abstract available. PMID 32717042
- [Background] Tipton KD, Hamilton DL, Gallagher IJ. Assessing the Role of Muscle Protein Breakdown in Response to Nutrition and Exercise in Humans. Sports Med. 2018 Mar;48(Suppl 1):53-64. doi: 10.1007/s40279-017-0845-5. PMID 29368185
- [Background] Kochlik B, Gerbracht C, Grune T, Weber D. The Influence of Dietary Habits and Meat Consumption on Plasma 3-Methylhistidine-A Potential Marker for Muscle Protein Turnover. Mol Nutr Food Res. 2018 May;62(9):e1701062. doi: 10.1002/mnfr.201701062. Epub 2018 Apr 19. PMID 29573154
- [Background] Peters NC, Contento IR, Kronenberg F, Coleton M. Adherence in a 1-year whole foods eating pattern intervention with healthy postmenopausal women. Public Health Nutr. 2014 Dec;17(12):2806-15. doi: 10.1017/S1368980014000044. PMID 24499772
- [Background] Sotos-Prieto M, Bhupathiraju SN, Mattei J, Fung TT, Li Y, Pan A, Willett WC, Rimm EB, Hu FB. Association of Changes in Diet Quality with Total and Cause-Specific Mortality. N Engl J Med. 2017 Jul 13;377(2):143-153. doi: 10.1056/NEJMoa1613502. PMID 28700845
- [Background] Milosevic I, Levy HC, Alcolado GM, Radomsky AS. The Treatment Acceptability/Adherence Scale: Moving Beyond the Assessment of Treatment Effectiveness. Cogn Behav Ther. 2015;44(6):456-69. doi: 10.1080/16506073.2015.1053407. Epub 2015 Jun 19. PMID 26091250
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Background] van der Wardt V, Harrison JK, Welsh T, Conroy S, Gladman J. Withdrawal of antihypertensive medication: a systematic review. J Hypertens. 2017 Sep;35(9):1742-1749. doi: 10.1097/HJH.0000000000001405. PMID 28486271
- [Derived] Zeiler E, Gabriel S, Ncube M, Thompson N, Newmire D, Scharf EL, Goldhamer AC, Myers TR. Prolonged Water-Only Fasting Followed by a Whole-Plant-Food Diet Is a Potential Long-Term Management Strategy for Hypertension and Obesity. Nutrients. 2024 Nov 20;16(22):3959. doi: 10.3390/nu16223959. PMID 39599745